CLINICAL TRIAL: NCT03907137
Title: Utilisation of Benralizumab in the Clinical Practise in Severe Eosinophilic Asthma Patients in Switzerland
Brief Title: Real World Study With Benralizumab in Severe Asthma in Switzerland
Acronym: BEEPS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00048
Record Dates: First submitted 2019-03-14; First posted 2019-04-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BEEPS describes the utility of patient reported outcomes (PRO) as simple, pragmatic, and sensitive tool to assess early treatment response of benralizumab to document the level of asthma control and change in medication after 1 to 16 weeks post-treatment initiation including use of OCS. The generated data on the time of asthma symptom relief after initiation of benralizumab will support patient management for a better disease control in severe asthma patients under benralizumab treatment. To assess long term outcomes the patients will have a last mandatory visit after 56 weeks, with no visits scheduled between week 16 and 56.

DETAILED DESCRIPTION:
The aim and objective of this single arm, prospective observational study is to describe patient reported outcomes (PRO) in severe eosinophilic asthma patients who are treated with benralizumab according to the label granted in Switzerland. The PRO measures consist of the weekly Asthma Control Questionnaire (ACQ-5) as well as Patient Global Impression of Change and Severity (PGI-C and PGI-S) collected at each visit (0, 1, 2, 4, 8, 16, 56 weeks). In addition the patient fills out twice daily the patient electronic asthma diary (eDiary) capturing daily symptoms and symptom free days together with a PEF (Peak Expiratory Flow) measurement. Persistance with eDiary and PEF will be assessed after 56 weeks. The percentage of patients successfully reducing their OCS dose will be evaluated after 16 weeks of treatment with benralizumab and if OCS reduction is persistent until week 56. Furthermore, the proportion of patients with an ACQ-5 score improvement of ≥ 0.5 after 8 weeks of treatment with benralizumab will be determined. In addition, the study will assess changes in FEV1 and FVC after 8, 16 and 56 weeks of treatment with benralizumab and describe retrospectively asthma disease history, past treatment status and current medication at baseline.

ELIGIBILITY:
Inclusion Criteria:

Subject eligible for enrolment in the study and treatment for benralizumab according to the specific Swiss label must meet all the following criteria:

1. Male or female patients older than 18 years with physician's confirmed diagnosis of severe, uncontrolled asthma according to ATS/ERS guidelines.
2. Asthma requiring high-dose ICS plus LABA as maintenance treatment.
3. Minimum of 2 exacerbations in the last 12 months.
4. Documented peripheral blood eosinophil count ≥ 300 cells/μL blood.
5. Provision of signed written informed consent form (ICF) indicating that they understand the purpose of the study and procedures required for participation in the study.
6. Patients must be able and willing to read and comprehend written instructions, and comprehend and complete the questionnaires required by the protocol (ACQ-5, PGI-C and PGI-S).

Exclusion Criteria:

Subjects meeting any of the following criteria will not be eligible to participate in the study:

1. Documented lung diseases other than asthma, e.g. COPD, and not within reimbursed label, e.g pregnancy or lactation.
2. Currently enrolled in an interventional clinical study in parallel, except:

   * Patients being in parallel documented in a national asthma registry.
   * Patients having completed any other clinical trial including those with biologic treatment.
3. An acute or chronic condition that, in the investigator's opinion, would limit the patients' ability to complete questionnaires or participate in this study or impact the interpretations of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit 77 male and female patients aged ≥ 18 years with severe, eosinophilic asthma who meet all inclusion criteria and none of the exclusion criteria. Approximately 15-20 specialist centres across Switzerland will participate in the study which have experience with biologic treatment, can initiate treatment with benralizumab and have a good oversight on the severe asthma population, as in some settings the patients are referred for longer term stationary care to achieve asthma control.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline ACQ-5 score after 8 weeks after initiation of benralizumab | 8 weeks
  The ACQ-5 (Asthma Control Questionnaire - 5 questions) consists of 5 questions about the asthma symptoms in the last 7 days. Each question has a scale from 0 (no symptoms) to 6 (most severe). The reported mean score of all questions describes the level of asthma control (0-6) whereby a mean score >1,5 is considered as uncontrolled asthma.

SECONDARY OUTCOMES:
Percentage of patients on OCS who were able to reduce their OCS after 16 weeks. | 16, 56 weeks
  In patients who take continuous oral corticosteroids (OCS) the fraction of patients who reduced the dosage of OCS is assessed. Daily oral OCS dosage in this patient group usually ranges from 2,5 to 40mg.
Change from baseline in ACQ 5 score up to 16 weeks after initiation of treatment with benralizumab. | 1, 2, 4, 16, 56 weeks
  The ACQ-5 (Asthma Control Questionnaire - 5 questions) consists of 5 questions about the asthma symptoms in the last 7 days. Each question has a scale from 0 (no symptoms) to 6 (most severe). The reported mean score of all questions describes the level of asthma control (0-6) whereby a mean score >1,5 is considered as uncontrolled asthma.
Proportion of patients with a total score improvement of ≥ 0.5 in ACQ-5 under treatment with benralizumab. | 1,2,4,8,16,56 weeks
  The ACQ-5 (Asthma Control Questionnaire - 5 questions) consists of 5 questions about the asthma symptoms in the last 7 days. Each question has a scale from 0 (no symptoms) to 6 (most severe). The reported mean score of all questions describes the level of asthma control (0-6) whereby a mean score >1,5 is considered as uncontrolled asthma.
Change from baseline in PGI-C in asthma. | 1, 2, 4, 8, 16, 56 weeks
  The Patient Global Impression of Change (PGI-C) rates the patients general impression of his asthma health status since study start on a scale from 1 to 7. 1 meaning much better, 4 equal and 7 much worse.
Change from baseline in PGI-S in asthma | 1, 2, 4, 8, 16, 56 weeks
  The Patient Global Impression of Severity (PGI-S) rates the current asthma status on a scale from 1 to 6. 1 meaning no symptoms and 6 meaning very heavy symptoms.
Asthma disease history | Baseline
  The time and age of first asthma diagnosis, the presence of allergic cofactors and the history of exacerbations in the last 12 month since study start will be recorded.
Past treatment status | Baseline
  Prescribed medication for Astma in the last 12 month before study enrollment will be recorded. Special emphasis will be put on inhallation therapy and OCS use and any changes. Any previous biological therapy will be recorded as well.
Patient demographics | Baseline
  Age (Years), sex (m/f), weight (kg) and height (cm) will be recorded

OTHER OUTCOMES:
Changes in PEF under treatment with benralizumab | 1, 2, 4, 8, 16, 56 weeks
  PEF=Peak Expiratory Flow; Measured in litres (l)
Outcome deterioration of asthma status (CompEx) with an electronic diary (app on smartphone) filled out by the patient. | Twice Daily throughout the study duration (16 weeks)
  The morning diary comprises four questions, the evening diary comprises three questions assessing the current asthma status.
  The scores will be summarised to defie a Compex event which is defined as 2 of the following criteria for ≥ 2 consecutive days:
  • ≥15% decrease from baseline in morning or evening PEF
  And at least one of the following:
  * ≥1.5 puffs increase from baseline in rescue medication morning or evening
  * ≥1 score increase from baseline, or the absolute maximal asthma symptom score in the morning or evening.
  Or one of the criteria above together with all diary variable showing a slope of worsening over at least a 5-day period.
Pre- and postbronchodilator changes in FEV1 under treatment with benralizumab. | 0, 8, 16, 56 weeks
  Forced Expiratory Volume in One Second (FEV1) is assessed by standard spirometry (measured in litres).
Pre- and postbronchodilator changes in FVC under treatment with benralizumab | 0, 8, 16, 56 weeks
  Forced vital capacity will be assessed by standard routine spirometry (measured in liters).
Change in OCS medication (median change in mg) | 4, 8, 16, 56 weeks
  Median OCS dose reduction
Percentage of patients with OCS reduction | 4, 8, 16, 56 weeks
  Proportion of patients with a ≥25%, ≥50%, ≥75% and 100% OCS dose reduction Percentage of patients on OCS who were able to reduce their OCS dose
Change of nasal polyposis relevant health status (taste and smell) | 1, 2, 4, 8, 16, 56 weeks
  For patients with nasal polyposis at baseline any improvement on taste/smell will be recorded categorically (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rothe, Dr. med., Principal Investigator — Kantonsspital Graubünden
Locations (10):
- Switzerland (10):
  - Research Site, Aathal
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Chur
  - Research Site, Geneva
  - Research Site, Liestal
  - Research Site, Lucerne
  - Research Site, Sion
  - Research Site, Wetzikon
  - Research Site, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: D3250R00048_BEEPS_CSR_Synopsis_022024_Redacted.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00048&attachmentIdentifier=a9bd9b0a-fb8d-46c4-98c4-58e1cb46f136&fileName=D3250R00048_BEEPS_CSR_Synopsis_022024_Redacted.pdf&versionIdentifier=